CLINICAL TRIAL: NCT07271160
Title: The Effect of Aromatherapy Foot Massage on Neuropathic Pain in Patients With Type2 Diabetes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Özlem Ceyhan, associate professor, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: aromatherapy foot massage
Record Dates: First submitted 2025-02-27; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes Mellitus (T2DM); Neuropathic Pain
Keywords: neuropathic pain; type 2 diabetes; aromatherapic massage
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Neuralgia | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Patients in the Intervention I group will receive aromatherapy foot massage. Patients in the Intervention II group will receive massage with sesame oil. The control group will not receive any application other than treatments.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- aromatherapy foot massage (Experimental): 'Patient Introduction Form', "DN4 neuropathic pain questionnaire", "Mcgill pain questionnaire short form" and "Pain-Activity Patterns scale" will be applied through face-to-face interview and the first aromatherapy foot massage will be applied when the patients in the intervention I group first arrive. Patients will be asked to massage the right foot for five minutes and the left foot for five minutes for a total of ten minutes before going to bed three days a week (Monday-Wednesday-Friday) in accordance with the foot massage application protocol.
  The 'Mcgill pain questionnaire short form' will be administered to the patients every week on Saturday at the same time by telephone. At the end of the fourth week, 'DN4 neuropathic pain questionnaire', 'Mcgill pain questionnaire short form' and 'Pain-Activity Patterns scale' will be applied again by telephone or face-to-face interview.
  Interventions: Other: intervention I group
- foot massage (Experimental): When the patients in the Intervention II group first arrive, the 'Patient Introduction Form', 'DN4 neuropathic pain questionnaire', 'Mcgill pain questionnaire short form' and 'Pain-Activity Patterns scale' will be applied through face-to-face interview and the first foot massage with sesame oil will be applied. Patients will be asked to massage the right foot for five minutes and the left foot for five minutes for a total of ten minutes before going to bed three days a week (Monday-Wednesday-Friday) in accordance with the foot massage application protocol.
  The 'Mcgill pain questionnaire short form' will be administered to the patients every week on Saturday at the same time by telephone. At the end of the fourth week, 'DN4 neuropathic pain questionnaire', 'Mcgill pain questionnaire short form' and 'Pain-Activity Patterns scale' will be applied again by telephone or face-to-face interview.
  Interventions: Other: Intervention II group
- Control Group (No Intervention): No application will be made to the control group, 'Patient Introduction Form', 'DN4 neuropathic pain questionnaire', 'Mcgill pain questionnaire short form' and 'Pain-Activity Patterns scale' will be collected by face-to-face interview.
  'Mcgill pain questionnaire short form' will be administered to the patients every week on Saturday at the same time by telephone. At the end of the fourth week, 'DN4 neuropathic pain questionnaire', 'Mcgill pain questionnaire short form' and 'Pain-Activity Patterns scale' will be applied again by telephone or face-to-face interview.

INTERVENTIONS:
Other: intervention I group — 'Patient Introduction Form', 'DN4 neuropathic pain questionnaire', 'Mcgill pain questionnaire short form' and 'Pain-Activity Patterns Scale' will be applied through face-to-face interview and the first aromatherapy foot massage will be applied when the patients in the intervention I group first arrive. Patients will be asked to massage their right foot for five minutes and their left foot for five minutes before going to bed three days a week (Monday-Wednesday-Friday) for a total of ten minutes in accordance with the foot massage application protocol. 'Mcgill pain questionnaire short form' will be administered to the patients every week on Saturday at the same time by telephone. At the end of the fourth week, 'DN4 neuropathic pain questionnaire', 'Mcgill pain questionnaire short form' and 'Pain-Activity Patterns Scale' will be administered again by telephone or face-to-face interview.
  Other Names: intervention II group
  Arms: aromatherapy foot massage
Other: Intervention II group — When the patients in the Intervention II group first arrive, the 'Patient Introduction Form', 'DN4 neuropathic pain questionnaire', 'Mcgill pain questionnaire short form' and 'Pain-Activity Patterns Scale' will be applied through face-to-face interview and the first foot massage with sesame oil will be applied. Patients will be asked to massage their right foot for five minutes and their left foot for five minutes before going to bed three days a week (Monday-Wednesday-Friday) for a total of ten minutes in accordance with the foot massage application protocol. 'Mcgill pain questionnaire short form' will be administered to the patients every week on Saturday at the same time by telephone. At the end of the fourth week, 'DN4 neuropathic pain questionnaire', 'Mcgill pain questionnaire short form' and 'Pain-Activity Patterns Scale' will be administered again by telephone or face-to-face interview.
  Other Names: intervention II
  Arms: foot massage

SUMMARY:
The aim of this clinical trial is to learn about the effect of aromatherapy foot massage on neuropathic pain in patients with Type 2 diabetes. In addition, while determining the effect of aromatherapy foot massage on neuropathic pain; it was also aimed to find the source of the reduction in pain.

The main questions he aimed to answer are as follows:

Does aromatherapy foot massage have an effect on neuropathic pain in patients with type 2 diabetes? Does foot massage have an effect on neuropathic pain in patients with type 2 diabetes? The researchers will compare an oil without aromatherapy oil with a placebo group to see if aromatherapy foot massage reduces neuropathic pain.

Participants:

Participants will perform the massage treatment three times a week for 4 weeks. Participants will perform foot massage for 10 minutes, 5 minutes on each foot. Participants will be evaluated by calling once a week for 4 weeks.

DETAILED DESCRIPTION:
Up to half of diabetic patients suffer from a complication known as diabetic neuropathy, which affects both the autonomic and peripheral nervous systems, with particular damage to the lower extremities. Diabetic neuropathy affects the peripheral sensory nerve endings of the hands and lower extremities, causing pain, numbness, burning and tingling sensations. Symptoms such as pain and burning experienced by diabetics cause a decrease in quality of life. In addition, the risk of ulceration in the feet is more than 15% and the risk of amputation is 15 times higher than non-diabetic individuals. Although diabetic neuropathy is one of the most serious complications of diabetes, its treatment is symptomatic.

In the presence of pain, complementary and integrative therapies such as opioid and non-opioid drugs, surgical methods, manual therapies and various mind-body practices are applied. Massage, one of these methods, is performed by manipulation of the soft tissues of the body. However, massage has the advantages of being applicable to almost every part of the body, not requiring any special equipment and not causing any serious complications. Another method, aromatherapy, uses natural plant extracts known as essential oils to improve physical, mental and emotional health. These essential oils are extracted from various parts of plants, including flowers, leaves, stems, roots and fruits. Aromatherapy oils can be inhaled as inhalers or applied to the skin through massage, baths or compresses. Physiological and pathophysiological benefits of aromatherapy oils on the nervous system have also been supported by studies.

Diabetic neuropathic pain has been associated with mental comorbidity, sleep disorders, more diabetes complications and lower quality of life. Therefore, it is essential to effectively manage pain in diabetic neuropathy and improve the quality of life of the individual. In a study examining the effects of aromatherapy massage on neuropathic pain severity and quality of life; it was found that neuropathic pain scores and quality of life scores improved significantly in the intervention group compared to the control group. In this study, it was not specified whether the reduction in neuropathic pain was the result of massage therapy or a specific essential oil in the aromatherapy mixture, since no intervention was performed in the control group. In our study; while determining the effect of aromatherapy foot massage on neuropathic pain; it was aimed to find the source of the reduction in pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a Douleur neuropathic pain questionnaire score of 4 and above,
* 18 years and over,
* No psychiatric illness,
* Patients who are able to answer all the questions,
* Turkish-speaking patients.

Exclusion Criteria:

* Patients who cannot be contacted,
* Any limb, vascular problem or wound that prevents the application of foot massage,
* Thrombophlebitis, occlusive arterial disease, fever, etc. Those who are inconvenient to massage due to illness,
* Patients who refused to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
McGILL PAIN SURVEY SHORT FORM (SF-MPQ) | 4 weeks
  The scale, which was first developed by Melzack (1987) and validated in Turkish by Yakut et al. (2006), includes 15 descriptive word groups including the characteristics of pain. Eleven of them evaluate the sensory dimension of pain and four of them evaluate the perceptual dimension of pain. These descriptive words are graded on an intensity scale from 0 to 3 (0 = none, 1 = mild, 2 = moderate, 3 = severe). In the first part of the scale, a total of three pain scores are obtained: sensory pain score, perceptual pain score and total pain score. Sensory pain score is between 0-33, perceptual pain score is between 0-12 and total pain score is between 0-45. An increase in the score indicates an increase in pain.

SECONDARY OUTCOMES:
DOULEUR NEUROPATHIC PAIN QUESTIONNAIRE (DN4) | The scale will be applied at the first match and at the end of the 4th week.
  The scale, which was developed by a French expert group (2005) and validated by Ünal Çevik et al. (2010) in Turkish, consists of 10 items. The first 7 items are related to pain characteristics and sensations and the remaining 3 items are related to examination. A score of '1' is given if the answer is 'yes' and '0' if the answer is 'no'. If the sum of all 10 items is calculated as 4 or more, the patient is defined as having neuropathic pain.

OTHER OUTCOMES:
PAIN-ACTIVITY PATTERNS SCALE (POAM-P/ AAPÖ) | The scale will be applied at the first match and at the end of the 4th week.
  The scale, which was first developed by Cane et al. (2013) and the Turkish validity and reliability of which was performed by Emine Tunç Süygün (2019), consists of 3 subgroups, namely avoidance, overdoing, and regularisation, and a total of 30 questions, 10 for each subgroup. In the scale, 'Individuals with chronic pain use different ways to do their daily activities. Think about how you usually do your daily activities. For each of the following statements, circle the numbers between 0 and 4 that best describe how you usually do your daily activities'. In answering the scale, a 5-point Likert scoring system is used, 0-never 2-sometimes 4-always. For the sub-groups of avoidance, overdoing and regularisation, the answers given to the questions belonging to the groups are summed separately and the participant's 3 separate sub-group scores are obtained. The total scores calculated for the subgroups vary between 0-40 points separately.

CONTACTS AND LOCATIONS:
Overall Officials: Özlem Ceyhan, Associate Professor, Study Director — TC Erciyes University
Locations (1):
- Nevsehir State Hospital, Nevşehir, Nevşehir Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
individual patient data will only be used within the scope of the study.

REFERENCES:
- [Background] Sattayakhom A, Wichit S, Koomhin P. The Effects of Essential Oils on the Nervous System: A Scoping Review. Molecules. 2023 Apr 27;28(9):3771. doi: 10.3390/molecules28093771. PMID 37175176
- [Background] Naranjo C, Ortega-Jimenez P, Del Reguero L, Moratalla G, Failde I. Relationship between diabetic neuropathic pain and comorbidity. Their impact on pain intensity, diabetes complications and quality of life in patients with type-2 diabetes mellitus. Diabetes Res Clin Pract. 2020 Jul;165:108236. doi: 10.1016/j.diabres.2020.108236. Epub 2020 May 26. PMID 32470476
- [Result] Rivaz M, Rahpeima M, Khademian Z, Dabbaghmanesh MH. The effects of aromatherapy massage with lavender essential oil on neuropathic pain and quality of life in diabetic patients: A randomized clinical trial. Complement Ther Clin Pract. 2021 Aug;44:101430. doi: 10.1016/j.ctcp.2021.101430. Epub 2021 Jun 18. PMID 34217127
- [Result] Gok Metin Z, Arikan Donmez A, Izgu N, Ozdemir L, Arslan IE. Aromatherapy Massage for Neuropathic Pain and Quality of Life in Diabetic Patients. J Nurs Scholarsh. 2017 Jul;49(4):379-388. doi: 10.1111/jnu.12300. Epub 2017 Jun 12. PMID 28605119
- See also: National Center for Complementary and Integrative Health — https://www.nccih.nih.gov/health/aromatherapy